CLINICAL TRIAL: NCT05651906
Title: The Role of Endothelial Glycocalyx in Kidney Transplantation
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Navrátil, MUDr., FEBU, Principal Investigator, Charles University, Czech Republic
Other Study IDs: GCX-KTX
Record Dates: First submitted 2022-11-14; First posted 2022-12-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplantation
Keywords: Endothelial; Glycocalyx
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donors
- Recipients
  Interventions: Procedure: Kidney Transplantation

INTERVENTIONS:
Procedure: Kidney Transplantation — Kidney transplantation as the best option for patients with end-stage kidney disease.
  Groups: Recipients

SUMMARY:
The goal of this observational study is detailed examination of endothelial glycocalyx in kidney transplantation. Researchers will evaluate markers of degradation of EG in blood and urine; and also perform direct visualisation of EG with sidestream dark field imaging (SDF) in both donors and recipients of kidney transplantation.

The aim is to summarize the current knowledge and to point out the importance of EG in kidney transplantation.

DETAILED DESCRIPTION:
The endothelial glycocalyx (EG) is a thin layer on the surface of the endothelium that plays an important role for microcirculation and tissue metabolism. The role of EG is diverse - it acts as a protection of the endothelium against shear stress which is mediated on the intracellular structures of endothelial cells, allows the interaction of blood elements and endothelium, prevents the formation of uncontrolled thrombosis and excessive oxidative stress by free radicals. EG dysfunction can occur with partial or complete loss of its components, resulting in impaired vascular regulation and increased vascular permeability. Disruption or dysfunction of EG has been associated with disease states such as diabetes, chronic kidney disease, inflammatory conditions, sepsis, hypernatraemia, hypervolaemia and ischaemia/reperfusion injury. Enzymes such as hyaluronidase and metalloproteinases can degrade the components of EG. Damage to EG leads to the release of breakdown products into the bloodstream which can be detected. There are also direct methods of visualization of EG. Thanks to advances in the study of EG in kidney transplantation a comprehensive relationship in this field and specific clinical aspects can be assessed. In the future exploring potential therapeutic options to protect EG may have implications for better graft function and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing kidney transplantation

Exclusion Criteria:

* Patients who don't sign the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group 1: Donors after brain death, Donors after circulatory death Group 2: Patients with end-stage renal disease who are eligible for kidney transplantation
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Examination of Endothelial Glycocalyx in Donors | 1 year
  Correlation between the status of EG in donors and kidney function after kidney transplantation (
Examination of Endothelial Glycocalyx in Recipients | 1 year
  Description of microcirculation directly from the kidney's surface in 1 and 20 minutes after reperfusion (with Side stream darkfield imaging and Perfused boundary region)

SECONDARY OUTCOMES:
Endothelial Glycocalyx under different settings | 1 year
  Description of EG in living donors, donors after brain death, donors after circulatory death (measurements of degradation products od EG - mainly syndecan-1 in blood and urine)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czech Republic, Czechia